CLINICAL TRIAL: NCT07131059
Title: MRD-positive AML: a Prospective, Single-arm, Multicenter Platform Clinical Study
Brief Title: MRD-positive AML Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024032
Record Dates: First submitted 2024-05-12; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-05

CONDITIONS: AML, Adult
Keywords: Measurable Residual Disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual | interventions — ivosidenib; gilteritinib; venetoclax; avapritinib; Daunorubicin; Cytarabine; Idarubicin; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- With lDH1 gene mutation (Experimental): Ivosidenib 500mg/d d1-28 ；Azacitidine 75mg/m2/d d1-7；Venetoclax400mg/d:d1-28
  Interventions: Drug: Ivosidenib; Drug: Venetoclax
- FLT3 gene mutation (Experimental): Gilteritinilb 120mg/d, d1 -28； Venetocax 400mg/d d1-28 400mg
  Interventions: Drug: Gilteritinib; Drug: Venetoclax
- NPM1 mutation or IDH2 mutation (Experimental): Azacitidine 75mg/m2/d d1-7；Venetoclax400mg/d d1-21 or Cytarabine 20mg/m2/d d1-10；Venetoclax 600mg/d d1-21
  Interventions: Drug: Venetoclax
- c-kit mutation (Experimental): Avapritinib 200mg/ day, 28 days a course
  Interventions: Drug: Avapritinib
- Daunorubicin/MTZ/Idarubicin+Cytarabine +Venetoclax (Experimental): Cytarabine 100mg/m2/d, d1-5； Daunorubicin 45mg/m2/d，d1-2；or Idarubicin 10mg/ m2/d，d1-2；or MTZ 8mg/ m2/d d1-2; Venetoclax 400mg d1-7
  Interventions: Drug: Venetoclax; Drug: Daunorubicin; Drug: Cytarabine; Drug: Idarubicin; Drug: MTZ
- Cytarabine+HHT+Venetoclax (Experimental): Cytarabine 100mg/ m2/d, d1-5; HHT 2mg/ m2 d1-5; Venetoclax 400mg d1-7
  Interventions: Drug: Venetoclax; Drug: Cytarabine; Drug: HHT
- Venetoclax+Azacitidine/Venetoclax+Cytarabine (Experimental): Azacitidine75 mg/m2 day1-7；Venetoclax 400mg day1-21 or，Cytarabine 20mg/m2 /day，day1-10； Venetoclax 600mg day1-21
  Interventions: Drug: Venetoclax; Drug: Cytarabine; Drug: Azacitidine

INTERVENTIONS:
Drug: Ivosidenib — 500mg d1-28
  Arms: With lDH1 gene mutation
Drug: Gilteritinib — 120mg d1-28
  Arms: FLT3 gene mutation
Drug: Venetoclax — 400mg d1-21 ; 400mg d1-7;400mg d1-28; 600mg d1-21
  Arms: Cytarabine+HHT+Venetoclax; Daunorubicin/MTZ/Idarubicin+Cytarabine +Venetoclax; FLT3 gene mutation; NPM1 mutation or IDH2 mutation; Venetoclax+Azacitidine/Venetoclax+Cytarabine; With lDH1 gene mutation
Drug: Avapritinib — 200mg d1-28.
  Arms: c-kit mutation
Drug: Daunorubicin — 45mg/m2/d d1-2;
  Arms: Daunorubicin/MTZ/Idarubicin+Cytarabine +Venetoclax
Drug: Cytarabine — 100mg/m2/d d1-5
  Arms: Cytarabine+HHT+Venetoclax; Daunorubicin/MTZ/Idarubicin+Cytarabine +Venetoclax; Venetoclax+Azacitidine/Venetoclax+Cytarabine
Drug: Idarubicin — 10mg/m2/d d1-2
  Arms: Daunorubicin/MTZ/Idarubicin+Cytarabine +Venetoclax
Drug: MTZ — 8mg/m2/d d1-2
  Arms: Daunorubicin/MTZ/Idarubicin+Cytarabine +Venetoclax
Drug: HHT — 2mg/m2/d d1-5
  Arms: Cytarabine+HHT+Venetoclax
Drug: Azacitidine — 75mgd/m2 d1-7.
  Arms: Venetoclax+Azacitidine/Venetoclax+Cytarabine

SUMMARY:
This clinical trial is a platform-type clinical study intended to investigate the efficacy and safety of MRD-positive acute myeloid leukemia patients after comprehensive treatment, which includes but is not limited to the following drugs and protocols: Chemotherapy, small molecule targeted drugs, demethylation drugs, liposome drugs and the combination of these drugs to form a combination of treatment regimen, the specific treatment regimen will be updated according to the results of this trial and the latest research progress at home and abroad.

DETAILED DESCRIPTION:
Patients aged 14 years or older with diagnosed AML (non-M3) who have achieved complete remission in bone marrow morphology but are positive for minimal residual disease by flow cytometry or have the following genetic mutations that can be detected by PCR: NPM1 mutation, IDH1/2 mutation, DEK-NUP214 (DEK-CAN), RUNX1-RUNX1T1(AML 1-ETO), or CBFβ-MYH 11[4]. NGS can detect mutations such as FLT3.

For eligible patients, the treatment plan is selected by the doctor in charge according to the specific conditions of the patient. During the treatment, patients can have hematopoietic stem cell transplantation at any time.

This study compared relapse-free survival and overall survival of MRD-positive patients after effective and persistent MRD treatment, and based on the results, observed the efficacy and safety of different treatment regiments for MRD-positive AML patients.

ELIGIBILITY:
Inclusion Criteria:

* AML (non-M3) compliant with WHO (2016) standards;
* In morphological complete remission.
* Mrd-positive patients: including bone marrow flow cytometry, PCR quantification of NPM1 mutations, PCR quantification of fusion genes (RUNX 1-RUNX1T1, CBFB-MYH11 and DEK-NUP214), or NGS detection of FLT3 mutation positive.
* Age over 14 years old, male or female. Informed consent must be signed prior to the commencement of all specific study procedures, and for those 14 years of age and older, informed consent must be signed by the patient or an immediate family member. Considering the patient's condition, if the patient's signature is not conducive to the treatment of the condition, the informed consent shall be signed by the legal guardian or the patient's immediate family.

Exclusion Criteria:

* Patients who intend to undergo hematopoietic stem cell transplantation within 4 weeks
* The diagnosis is APL
* Those who were not considered suitable for inclusion by the researchers.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-11 (Actual); Primary Completion 2026-05-10 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
relapse-free survival rate | up to 6 months

SECONDARY OUTCOMES:
Measurable Residual Disease | up to 6 months
Proportion of MRD turning negative | up to 6 months
Overall survival(OS ) rate | From the time the patients participated in the clinical trial until the patient died
Cumulative relapse rate | From the time the patients participated in the clinical trial until the patient relapsed
Adverse Events (AEs) | up to 2 years
The incidence of adverse events such as serious infections during treatment | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Huui Wei, doctor, Principal Investigator — Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No